CLINICAL TRIAL: NCT02602574
Title: Endoscopic Retrograde Cholangiopancreatography (ERCP)-Induced and Non-ERCP Induced Acute Pancreatitis: Two Distinct Clinical and Immunological Entities?
Brief Title: ERCP-induced and Non-ERCP Induced Acute Pancreatitis: Two Distinct Clinical and Immunological Entities?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Goran Hauser, doc.dr.sc. Goran Hauser, dr. med., University Hospital Rijeka
Other Study IDs: PEP 2015
Record Dates: First submitted 2015-10-29; First posted 2015-11-11 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Pancreatitis; Heat-Shock Proteins; Pentraxin 3 protein; C-Reactive Protein; procalcitonin; Interleukin-1 beta; Leukocytes, Mononuclear; Killer Cells, Natural; natural-killer group 2, member D receptor
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, mononuclear cell suspension
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ERCP- induced acute pancreatitis: All patients with indication for ERCP will be prepared for ERCP. One hour before and 4-6 hours after the procedure 10 mL of blood sample and urine sample will be collected.
  24 hours after the procedure all patients will be taken 30 ml of heparinized peripheral venous blood and urine sample.
  Upon clinical and laboratory confirmation of acute pancreatitis according to ESGE guidelines for post-ERCP pancreatitis, will be further monitored during hospitalization for evaluation of the severity of the disease.
  Interventions: Other: heparinized peripheral venous blood and urine sample.
- non -ERCP acute pancreatitis: All patients with acute pancreatitis according to Atlanta criteria admitted through Emergency Department will be taken 30 ml of heparinized peripheral venous blood and urine sample upon 24 hours after the clinical symptoms have started. 10 mL of collected blood samples will be examined in the Department of Laboratory Medicine. Other 20 mL of blood samples will be sent to Department of Physiology and Immunology, School of Medicine where immunologic analysis will be performed.
  This group of patients will be further monitored during hospitalization for evaluation of the severity of the disease. Severity of the disease will be assessed according to the Atlanta criteria.
  Interventions: Other: heparinized peripheral venous blood and urine sample.
- Control group: Control group will consist of patients who underwent ERCP but didn't develop acute pancreatitis. One hour before and 4-6 hours after the procedure 10 mL of blood sample and urine sample will be collected.
  24 hours after the procedure all patients will be taken 30 ml of heparinized peripheral venous blood and urine sample.
  Interventions: Other: heparinized peripheral venous blood and urine sample.

INTERVENTIONS:
Other: heparinized peripheral venous blood and urine sample. — All patients will be taken heparinized peripheral venous blood and urine sample

SUMMARY:
Post endoscopic pancreatitis (PEP) has different initial immunologic response to primary injury compared to acute pancreatitis of other etiology (non-PEP AP).

The purpose of this study is to compare initial immunologic response, 24 h after primary injury, in patients with PEP and patients with acute pancreatitis of other etiology.

DETAILED DESCRIPTION:
PROTOCOL:

All patients with indication for endoscopic retrograde cholangiopancreatography (ERCP) will be prepared for ERCP on the following protocol: they will be instructed not to eat 4 to 6 hours before the procedure. Immediately before the procedure they will be administrated with Diclophenac Sodium 100 mg suppositories. One hour before the procedure 10 mL of blood sample and urine sample will be taken and analyzed in laboratory premises incorporated in University Hospital Centre Rijeka for following parameters: values of amylase in serum and urine and lipase in serum, liver enzyme tests and kidney function. 4-6 hours after ERCP is performed, 10 mL of blood sample will be taken and analyzed in laboratory premises incorporated in University Hospital Centre Rijeka for following parameters: values of amylase in serum and urine and lipase in serum, liver enzyme tests and kidney function.

24 hours after the procedure all patients will be taken 30 ml of heparinized peripheral venous blood and urine sample. 10 mL will be examined in the Department of Laboratory Medicine, Clinical Hospital Centre for following parameters: values of amylase in serum and urine and lipase in serum, liver enzyme tests and kidney function. Urine sample collected after the procedure will be used to evaluate amylase levels. Other 20 mL of blood samples will be sent to Department of Physiology and Immunology, School of Medicine where immunologic analysis will be performed. All patients who underwent ERCP will be divided into two groups. First group (PEP group) will be made of patients who developed acute pancreatitis following ERCP. Upon clinical and laboratory confirmation of acute pancreatitis according to European Society of Gastrointestinal Endoscopy (ESGE) guidelines for post-ERCP pancreatitis, will be further monitored during hospitalization for evaluation of the severity of the disease. Severity of the disease will be assessed according to the Cotton criteria for the severity of post-ERCP pancreatitis. Group of patients who underwent ERCP but didn't develop acute pancreatitis within 24 hours after the procedure, according to ESGE guidelines will be used as a control group (non-PEP group).

All patients with acute pancreatitis according to Atlanta criteria admitted through Emergency Department will be taken 30 ml of heparinized peripheral venous blood and urine sample upon 24 hours after the clinical symptoms have started (upper abdominal pain often radiating through to the back). 10 mL of collected blood samples will be examined in the Department of Laboratory Medicine, Clinical Hospital Centre for following parameters: values of amylase in serum and urine and lipase in serum, liver enzyme tests and kidney function. Other 20 mL of blood samples will be sent to Department of Physiology and Immunology, School of Medicine where immunologic analysis will be performed. This group of patients will be further monitored during hospitalization for evaluation of the severity of the disease. Severity of the disease will be assessed according to the Atlanta criteria.

METHODS AND MATERIALS

Laboratory parameters

For each patient included in the study blood and urine analysis will be performed in the Department of Laboratory Medicine, Clinical Hospital Centre Rijeka. Basic hematology tests will include: total blood count - a count of the total number of red blood cells, white blood cells and platelets present in blood, values of hemoglobin and hematocrit. Biochemical analysis of blood serum will include: values of amylase and lipase in serum, sodium, potassium, glucose, liver enzymes (aspartate aminotransferase (AST), alanine aminotransferase (ALT), Gama-glutamyl transferase (GGT), alkaline phosphatase (ALP)) direct and indirect bilirubin, kidney function (serum urea and creatinine, estimated glomerular filtration (eGFR)), C-reactive protein and acid-base status of arterial blood.

Immunological methods

For each patient included in the study immunologic analysis of blood samples (24 hours after the procedure or onset of the symptoms) will be performed in Department of Physiology and Immunology, School of Medicine in Rijeka, Croatia.

Isolation of peripheral blood mononuclear cells Twenty milliliters of peripheral blood will be acquired in Vacutainer (Becton Dickinson, Franklin Lakes, NY), overlaid onto Lymphoprep (Nycomed Pharma AS, Oslo, Norway) and centrifuged (20 min at 600 g). After the centrifugation, the cells from the interface will be collected and washed twice in Roswell Park Memorial Institute (RPMI) 1640 medium (Auckland, NZ) and used immediately for further experimental procedure. The viability of the cells was >95% will be assessed with propidium iodide 0.5 mg/ml/106 cells (Sigma-Aldrich Chemie) and a flow cytometer (FACSCalibur, Becton Dickinson, San Jose, USA)

Detection of cell surface Peripheral blood mononuclear cells (PBMC) will be stained for 30 min at 40 degrees Celsius with different combinations of Phycoerythrin (PE) - Cyanine (Cy) anti-cluster of differentiation (CD) 3 monoclonal antibody (mouse Antibody (mAb), Immunoglobulin G 1 (IgG1)), PE-conjugated anti-cluster of differentiation (CD)56 mAb (mouse B159, IgG1) and fluorescein isothiocyanate (FITC)-conjugated anti-natural-killer group 2, member D (NKG2D) mAb (5C6). FITC-, PE- and PE-Cy conjugated mouse isotype match antibodies will be used to set negative controls for each class of antibody used.

Stained cell samples will be analyzed by flow cytometry using FACSCalibur flow cytometer (Becton Dickinson & Co, San Jose, USA).

Detection of cytokine Interleukin (IL)-1 beta (β) and heat shock protein (HSP) 70, 27.

For the quantitative determination of human IL-1 β concentrations in plasma,Human IL-1 ELISA (Enzyme-Linked Immunosorbent Assay) Kit will be used.

For the quantitative determination of heat shock protein (HSP) 70 and 27 in plasma, HSP 70 High sensitivity ELISA Kit and HSP 27 ELISA kit will be used.

Detection of pentraxin 3 (PTX 3) and procalcitonin For the quantitative determination of human pentraxin 3 (PTX) and procalcitonin concentrations in plasma specific ELISA Kit will be used.

ELIGIBILITY:
Inclusion Criteria:

* all patients underwent to ERCP irrespectively about the diagnosis
* all patients with diagnosed acute pancreatitis according to Atlanta criteria admitted through Emergency Department within 24 hours of onset of symptoms.

Exclusion Criteria:

* unwillingness or inability to consent for the study
* anticipated inability to follow protocol, previous ERCP, acute cholecystitis and/or cholangitis
* active or recent (within 4 weeks) gastrointestinal hemorrhage
* existing acute pancreatitis (lipase peak) within 72 hours prior to ERCP
* intrauterine pregnancy, breast feeding mother
* patients with chronic inflammatory diseases (e.g. IBD) systemic inflammatory and autoimmune disorders (e.g. systemic lupus erythematosus, ) or acute inflammatory diseases (e.g. pneumonia, pyelonephritis or sepsis of any cause)
* patients on immunomodulatory or immunosuppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with indication for ERCP and all patients with acute pancreatitis admitted through Emergency Department
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of initial immunologic response in patients with PEP and patients with AP of other etiology (Number of Participants With Abnormal Laboratory Values) | 24 hours after the primary injury
  Number of Participants With Abnormal Laboratory Values

SECONDARY OUTCOMES:
Correlation between differences in initial inflammatory response and clinical outcomes of AP (biliary and alcoholic) and PEP (Number of Participants With Abnormal Laboratory Values) | 1 month
  Number of Participants With Abnormal Laboratory Values

CONTACTS AND LOCATIONS:
Overall Officials: Davor Štimac, MD, PhD, Study Chair — Clinical Hospital Centre Rijeka
Locations (1):
- Clinical Hospital Centre, Rijeka, Kresimirova 42, Croatia

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Background] Kylanpaa L, Rakonczay Z Jr, O'Reilly DA. The clinical course of acute pancreatitis and the inflammatory mediators that drive it. Int J Inflam. 2012;2012:360685. doi: 10.1155/2012/360685. Epub 2012 Dec 12. PMID 23304633
- [Background] Demols A, Deviere J. New frontiers in the pharmacological prevention of post-ERCP pancreatitis: the cytokines. JOP. 2003 Jan;4(1):49-57. PMID 12555016
- [Background] Testoni PA, Vailati C, Giussani A, Notaristefano C, Mariani A. ERCP-induced and non-ERCP-induced acute pancreatitis: Two distinct clinical entities with different outcomes in mild and severe form? Dig Liver Dis. 2010 Aug;42(8):567-70. doi: 10.1016/j.dld.2009.10.008. Epub 2009 Dec 16. PMID 20018574
- [Background] Fung AS, Tsiotos GG, Sarr MG. ERCP-induced acute necrotizing pancreatitis: is it a more severe disease? Pancreas. 1997 Oct;15(3):217-21. doi: 10.1097/00006676-199710000-00001. PMID 9336783
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995